CLINICAL TRIAL: NCT03639051
Title: A Multicenter, Randomized, Sham-controlled Study to Evaluate Safety and Efficacy After Treatment with the Nuvaira™ Lung Denervation System in Patients with Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluation of the Safety and Efficacy of TLD in Patients with COPD
Acronym: AIRFLOW-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D0543
Record Dates: First submitted 2018-08-08; First posted 2018-08-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized with equal allocation (1:1) into two arms: TLD therapy plus optimal medical care (Active Treatment) and optimal medical care (Sham Control). Randomization of subjects will be stratified based on investigational site, participation in a pulmonary rehabilitation maintenance program and baseline use of an inhaled corticosteroid at the time of enrollment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject and assessor double-blinding will be maintained through 1 year post-procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): Target Lung Denervation (TLD) with the Nuvaira Lung Denervation System (RF energy delivered) and optimal medical care for COPD.
  Interventions: Device: Targeted Lung Denervation (TLD); Other: Optimal Medical Care
- Sham Control (Sham Comparator): Sham Targeted Lung Denervation (TLD) procedure with the Nuvaira Lung Denervation System (catheter placement and balloon deployment in all treatment locations, no RF energy delivered) and optimal medical care for COPD.
  Interventions: Other: Optimal Medical Care

INTERVENTIONS:
Device: Targeted Lung Denervation (TLD) — Targeted Lung Denervation (TLD) Therapy is a bronchoscopically guided, minimally invasive procedure using the Nuvaira™ Lung Denervation System.
  Other Names: TLD, TLD Therapy
  Arms: Active Treatment
Other: Optimal Medical Care — Taking regular maintenance medication that minimally includes a long-acting muscarinic antagonist (LAMA) and a long-acting beta2-agonist (LABA).

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of the Nuvaira Lung Denervation System (Nuvaira System) in the treatment of COPD.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the superiority of treatment with the Nuvaira Lung Denervation System (Active Treatment arm) compared to a sham procedure (Sham Control arm) to decrease moderate or severe exacerbations in subjects with COPD on optimal medical care.

The secondary objective is to compare long-term safety, and other efficacy assessments between the Active Treatment arm and the Sham Control arm.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥40 years of age at the time of consent;
* Women of child bearing potential must not be pregnant, evidenced by a negative pregnancy test (blood or urine) pre-treatment, or lactating and agree not to become pregnant for the duration of the study;
* Smoking history of at least 10 pack years;
* Not smoking or using any other inhaled substance (e.g., cigarettes, vaping, cannabis, pipes) for a minimum of 2 months prior to consent and agrees to not start for the duration of the study;
* Subject has received a flu vaccination within the 12 months prior to the procedure or agrees to obtain vaccination once it becomes available and agrees to annual vaccinations for the duration of the study;
* Resting SpO2 ≥89% on room air at the time of screening;
* CAT score ≥10 at the time of screening;
* Diagnosis of COPD with 25%≤ FEV1 ≤80% of predicted, PaCO2 ˂ 50 (if FEV1 ˂30%) and FEV1/FVC <70% (post-bronchodilator);
* Documented history of ≥ 2 moderate COPD exacerbations or ≥ 1 severe COPD exacerbation leading to hospitalization in the 12 months prior to consent with at least one exacerbation occurring while the subject was on optimal medical care (taking LAMA and a LABA, or scheduled SABA or SAMA instead of either a LAMA or LABA, not both, as regular respiratory maintenance medication);
* Subject is on optimal medical care at the time of consent;
* If subject has participated in a formal pulmonary rehabilitation program recently, program completion must have occurred ≥3 months prior to consent; if in a maintenance program, subject agrees to continue their current program through their 12-month follow-up visit;
* Subject is a candidate for bronchoscopy in the opinion of the physician or per hospital guidelines and is able to discontinue blood thinning medication peri-procedurally;
* The subject is able and agrees to complete all protocol required baseline and follow-up tests and assessments including taking certain medications (e.g., azithromycin, prednisolone/prednisone);
* Subject has provided written informed consent using a form that has been reviewed and approved by the Institutional Review Board (IRB)/Ethics Committee (EC).

Exclusion Criteria:

* Body Mass Index <18 or >35;
* Subject has an implantable electronic device and has not received appropriate medical clearance;
* Uncontrolled diabetes in the opinion of the investigator;
* Malignancy treated with radiation or chemotherapy within 1 year of consent;
* Asthma as defined by the current Global Initiative for Asthma (GINA) guidelines;
* Subject diagnosed with a dominant non-COPD lung disease or condition affecting the lungs, which is the main driver of the subjects clinical symptoms (e.g., cystic fibrosis, paradoxical vocal cord motion, eosinophilic granulomatosis with polyangiitis (EGPA), allergic bronchopulmonary aspergillosis, interstitial lung disease or active tuberculosis) or has a documented medical history of pneumothorax within 1 year of consent;
* Clinically relevant bronchiectasis, defined as severe single lobe or multilobar broncial wall thickening associated with airway dilation on CT scan leading to cough and tenacious sputum on most days;
* Pre-existing diagnosis of pulmonary hypertension, clinical evidence of pulmonary hypertension (e.g., cardiovascular function impairment including peripheral edema) and mPAP ≥25 mmHg at rest by right heart catheterization (or estimated right ventricular systolic pressure >50 mmHg by echocardiogram if no previous right heart catheterization);
* Myocardial infarction within last 6 months, EKG with evidence of life threatening arrhythmias or acute ischemia, pre-existing documented evidence of an LVEF <40%, stage C or D (ACC/AHA) or Class III or IV (NYHA) congestive heart failure, or any other past or present cardiac findings that make the subject an unacceptable candidate for a bronchoscopic procedure utilizing general anesthesia;
* Surgical procedure(s) on the stomach, esophagus or pancreas performed ≤2 years of consent or ongoing related symptoms within the past year;
* Symptomatic gastric motility disorder(s) (e.g., gastroparesis) as evidenced by a GCSI score ≥18.0, severe uncontrolled GERD (e.g., refractory heartburn, endoscopic esophagitis) or severe dysphagia (e.g., esophageal stricture, achalasia, esophageal spasm);
* Any disease or condition that might interfere with completion of a procedure or this study (e.g., structural esophageal disorder, life expectancy <3 years);
* Prior lung or chest procedure (e.g., lung transplant, LVRS, BLVR, lung implant, metal stent, valves, median sternotomy, bullectomy, lobectomy, segmentectomy or other interventional lung or chest procedure) performed ≤1 year of consent; NOTE: Any metal in the chest must be ≥5 cm away from the anticipated treatment location(s). Subjects with explanted lung valve(s) allowed if explant occurred ≥3 months prior to treatment.
* Daily use of >10 mg of prednisone or its equivalent at the time of consent;
* Chronic use of >40 mg MEDD opioid only medication per day;
* Known contraindication or allergy to medications required for bronchoscopy or general anesthesia (e.g., lidocaine, atropine, propofol, sevoflurane) that cannot be medically controlled;
* Baseline chest CT scan reveals bronchi anatomy cannot be fully treated with available catheter sizes, presence of severe emphysema >50%, lobar attenuation area or severe bullous disease (>1/3 hemithorax) (as determined by the CT core lab using a single density mask threshold of -950 HU) or discovery of a mass that requires treatment;
* Subject is currently enrolled in another interventional clinical trial that has not completed follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Moderate or severe COPD exacerbations | Randomization to 12 Months
  A COPD exacerbation will be defined as a complex of respiratory events/symptoms (increase or new onset) of more than one of the following: cough, sputum, wheezing, dyspnea or chest tightness with at least one symptom lasting three days requiring treatment with antibiotics and/or systemic steroids (moderate exacerbation) and/or hospital admission (severe exacerbation).

SECONDARY OUTCOMES:
Time to first severe COPD exacerbation | Randomization to 12 Months
  Defined as a comparison between study arms of the survival distributions for events based on log-rank tests
Time to first severe COPD exacerbation (Subgroup) | Randomization to 12 months
  Defined as a comparison between study arms of the survival distributions for events based on log-rank tests, only for the subgroup of subjects who had a severe COPD exacerbation in the year prior to randomization.
Change in St. George's Respiratory Questionnaire COPD Version (SGRQ-C) Total score | Randomization to 12 months
  Defined as a comparison between study arms of the mean change in FVC based on a linear model for change in SGRQ-C, adjusted for baseline SGRQ-C.
  The SGRQ-C is a disease-specific HRQL questionnaire with a total and three component scores for: symptoms, activity and impacts; each score ranges from 0 (no impairment) to 100 (worst possible). A difference in four units in the SGRQ-C score is considered the minimum clinically important difference (MCID).
Change in FVC | Randomization to 12 Months
  Defined as a comparision between study arms of the mean change in FVC based on a linear model for change in FVC, adjusted for baseline FVC.
Change in FEV1 | Randomization to 12 months
  Defined as a comparison between study arms of the mean change in FEV1 based on a linear model for change in FEV1, adjusted for baseline FEV1.
Transition Dyspnea Index (TDI) | Randomization to 12 months
  Defined as a comparison between study arms of the TDI based on a linear model for change in TDI.
Change in RV | Randomization to 12 months
  Defined as a comparison between study arms of the mean change in RV based on a linear model for change in RV, adjusted for baseline RV.
Time to first respiratory-related hospitalization | Randomization to 12 Months
  Defined as a comparison between study arms of the survival distributions for events based on log-rank tests.
Change in Short Form Health Survey (SF-36) total score | Randomization to 12 Months
  Defined as a comparison between study arms of the mean change in SF-36 total score based on a linear model for change in SF-36 total score, adjusted for baseline SF-36 total score.
  SF-36 is composed of eight multi-item scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health), with scores for each of these scales (or dimensions) ranging from 0 to 100. Higher scores indicate higher HRQoL.
CAT responders | Randomization to 12 Months
  Defined as a comparison between study arms of the proportion of subjects with a greater than or equal to 2 point decrease in CAT.
  The CAT is a disease-specific HRQL with eight questions; each score ranges from 0 (no impairment) to 5 (worst possible). The CAT has a scoring range of 0-40. Higher scores denote a more severe impact of COPD on a patient's life. A difference in 2 units in the CAT score over 2 to 3 months suggests a clinically significant difference or change in health status.

OTHER OUTCOMES:
Changes in quality of life | Randomization to 6, 12 Months
  Change in St. George's Respiratory Questionnaire (SGRQ-C), COPD Assessment Test (CAT) and Short Health Survey (SF-36) scores
Adverse event rates | Randomization to 12 Months, 3 to 12 Months
  Defined as the total number of events per total number of treatment years including moderate or severe COPD exacerbations, severe COPD exacerbations, respiratory-related hospitalizations, and lower respiratory-related adverse events
Time to first event | 3 to 12 Months
  Defined as comparison between study arms of the survival distributions for events based on log-rank tests including moderate or severe COPD exacerbations, severe exacerbations and respiratory-related hospitalizations
Changes in lung function | Randomization to 12 Months
  Changes in Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC) and Body plethysmography measures (IC, TLC, RV)
Changes in dyspnea | Randomization to 12 Months
  Changes in dyspnea including Modified Medical Research Council (mMRC) Dyspnea Scale scores and Baseline and Transition Dyspnea Indexes (BDI/TDI) scores
Healthcare utilization | Randomization to 12 Months
  Defined as respiratory-related unscheduled clinic visits, ER visits and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sciurba, MD, Principal Investigator — University of Pittsburgh Medical Center; Dirk-Jan Slebos, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (33):
- United States (20):
  - University of Alabama at Birmingham (UAB) Lung Health Center, Birmingham, Alabama
  - HonorHealth, Phoenix, Arizona
  - UC Davis, Sacramento, California
  - Harbor UCLA, Torrance, California
  - Ascension St. Vincent's, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Suburban Lung Associates, Elk Grove Village, Illinois
  - University of Louisville, Louisville, Kentucky
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - First Health of the Carolinas, Pinehurst, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - St. Davids HealthCare, Georgetown, Texas
  - Houston Methodist Hospital, Houston, Texas
- Krankenhaus Nord - Klinik Floridsdorf, Vienna, Austria
- France (8):
  - CHU de Grenoble, Grenoble, Cedex 9
  - Hopital Larrey, Toulouse, Cedex 9
  - Hopital de la Cavale Blanche, Brest
  - Arnaud de Villeneuve Hospital, Montpellier
  - Hopital Pasteur, Nice
  - Bichat-Claude Bernard Hospital, Paris
  - CHU de Reims, Reims
  - CHU de Strasbourg, Strasbourg
- Thorax Klinik Heidelberg, Heidelberg, Germany
- Netherlands (2):
  - UMC, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
- Royal Brompton Harefield Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, ending 36 months following article publication.
Access Criteria: Researchers whose proposed use of the data has been approved by a review committee identified for this purpose will have access to the data required to achieve aims in the approved proposal. Proposals should be directed to pjohnson@nuvaira.com. (Link to be provided).

REFERENCES:
- [Derived] Shah PL, Slebos DJ, Sue R, Bhatt SP, Ghattas C, Strange C, Degano B, Valipour A, Eisenmann S, De Cardenas J, Marquette CH, Soto-Soto J, Sciurba FC, Conway F, Tonkin J, Tana A, Marchetti N, Hartman JE, Heluain V, Guibert N, Criner GJ. Randomized Sham-controlled Trial of Targeted Lung Denervation in Patients with Chronic Obstructive Pulmonary Disease (AIRFLOW-3). Am J Respir Crit Care Med. 2025 Dec;211(12):2318-2329. doi: 10.1164/rccm.202502-0404OC. PMID 40920914
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989
- [Derived] Slebos DJ, Degano B, Valipour A, Shah PL, Deslee G, Sciurba FC; AIRFLOW-3 Trial Study Group. Design for a multicenter, randomized, sham-controlled study to evaluate safety and efficacy after treatment with the Nuvaira(R) lung denervation system in subjects with chronic obstructive pulmonary disease (AIRFLOW-3). BMC Pulm Med. 2020 Feb 13;20(1):41. doi: 10.1186/s12890-020-1058-5. PMID 32054473